CLINICAL TRIAL: NCT00269594
Title: An Open-Label Study of Lamictal In Neurotic Excoriation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0510M77009
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2007-04-30 (Estimated); Status verified 2007-04

CONDITIONS: Neurotic Disorders; Obsessive-Compulsive Disorder
Keywords: Skin; Picking; Pick; Neurotic Excoriation
MeSH Terms: conditions — Neurotic Disorders; Obsessive-Compulsive Disorder | interventions — Lamotrigine

INTERVENTIONS:
Drug: Lamictal (lamotrigine)

SUMMARY:
The goal of the proposed study is to evaluate the efficacy and safety of Lamictal in neurotic excoriation. Twenty subjects with neurotic excoriation will receive 12 weeks of open-label treatment with Lamictal. The hypothesis to be tested is that Lamictal will be effective and well tolerated in patients with neurotic excoriation. The proposed study will provide needed data on the treatment of a disabling disorder that currently lacks a clearly effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* men and women age 18-65
* current diagnosis of neurotic excoriation

Exclusion Criteria:

* unstable medical illness or clinically significant abnormalities on prestudy laboratory tests or physical examination
* history of seizures
* myocardial infarction within 6 months
* current pregnancy or lactation, or inadequate contraception in women of childbearing potential
* a need for medication other than Lamictal with possible psychotropic effects or unfavorable interactions with Lamictal
* clinically significant suicidality
* lifetime history of DSM-IV bipolar disorder type I, dementia, or schizophrenia or any other DSM-IV psychotic disorder
* current or recent (past 3 months) DSM-IV substance abuse or dependence
* illegal substance use within 2 weeks of study initiation
* initiation of psychotherapy or behavior therapy from a mental health professional within 3 months prior to study baseline
* previous treatment with Lamictal
* treatment with investigational medication or depot neuroleptics within 3 months, with fluoxetine within 6 weeks, or with other psychotropics within 2 weeks prior to study baseline
* current treatment with an anti-epileptic medication and
* patients who have previously been diagnosed with a medical condition that cause skin itchiness (e.g. liver, kidney, and blood diseases, etopic allergies)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-01; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale Modified for Neurotic Excoriation

SECONDARY OUTCOMES:
Skin Picking Symptom Assessment Scale (SP-SAS) and the Clinical Global Impression scale

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, JD, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Grant JE, Odlaug BL, Kim SW. Lamotrigine treatment of pathologic skin picking: an open-label study. J Clin Psychiatry. 2007 Sep;68(9):1384-91. doi: 10.4088/jcp.v68n0909. PMID 17915977